CLINICAL TRIAL: NCT05530863
Title: Behavioral Relaxation Approaches for Insomnia in Pregnant Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Nalaka Gooneratne, Principal Investigator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 848419
Record Dates: First submitted 2022-03-24; First posted 2022-09-07 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Sleep Initiation and Maintenance Disorders; Pregnancy Related
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Hygiene (Active Comparator): This arm will receive behavioral education, such as sleep hygiene and other advice. Additional details cannot be provided since that will compromise the participant blinding
  Interventions: Behavioral: Sleep Hygiene
- ART and Sleep Hygiene (Experimental): This arm will receive behavioral education, such as sleep hygiene and other training. Additional details cannot be provided since that will compromise the participant blinding
  Interventions: Behavioral: Assisted Therapy; Behavioral: Sleep Hygiene

INTERVENTIONS:
Behavioral: Assisted Therapy — The participant will receive coaching calls and support
  Arms: ART and Sleep Hygiene
Behavioral: Sleep Hygiene — Standard Sleep Hygiene instructions.

SUMMARY:
This study will evaluate the effect of a simplified behavioral relaxation intervention to improve insomnia in pregnant women

DETAILED DESCRIPTION:
This is a randomized, 60-day research study that is evaluating the effect of a simplified behavioral relaxation intervention in pregnant and postpartum patients aimed to improve their insomnia symptoms. The investigators will be enrolling a total of 20 patients who indicate self-reported insomnia symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 55
* In second or third trimester of pregnancy (Gestation weeks 18-32)
* Able to speak, read and write fluent English
* Has regular access to a smartphone and/or smart tablet
* sleep onset latency (SOL) or nocturnal awakening need be 30 min or more for ≥3 nights/week, must persist for at least 1 month

Exclusion Criteria:

* Participants with fixed night shift work between midnight and 5 am, or rotating work schedules requiring night shifts during the study period.
* Medical or other factors that, in the opinion of the study research team, would interfere with their ability to participate in the intervention (such as inability to participate in the ART due to blindness)

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-09-27 (Estimated); Study Completion 2027-09-27 (Estimated)

PRIMARY OUTCOMES:
PSQI, Sleep Quality | 30 days
  Measured by a single item score, sleep quality is the measurement of how restful and restorative the sleep of an individual is. Pittsburgh Sleep Quality Index: Well- known questionnaire used to measure sleep quality in various patient groups. For overall sleep quality, the minimum score= 0 (better) and the maximum score=3 (worse).
Total Wake Time, Sleep Diary | 30 days
  A sleep diary will be used to gather information about the participants daily sleep pattern and schedule; gold standard of care for insomnia. This instrument will also be used to check adherence to the Gratification practice of the ART intervention. This will be administered during pre-screening and intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Nalaka Gooneratne, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No